CLINICAL TRIAL: NCT02369237
Title: A Non-invasive Device to Determine Iron Deficiency Anemia in Children of Different Age Groups With Renal Failure
Brief Title: Non-invasive Determination of Anemia in Children With Renal Failure
Status: Completed | Type: Observational
Sponsor: Center for Studies of Sensory Impairment, Aging and Metabolism (Other)
Collaborators: Hildegrad Grunow Foundation (Unknown); MBR Optical Systems (Unknown)
Responsible Party: Sponsor
Other Study IDs: CeSSIAM_03
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Anemia and inflammation are very common in patients with renal diseases. The most common procedure to detect anemia is to determine blood hemoglobin concentrations. The Haemospect® is a portable device for non-invasive hemoglobin determination that works with a sensor that is applicable in infants and adults alike.

The objective of this trial is to collect spectra with the non-invasive Haemospect® device in children of different age groups with renal failure and different hemoglobin concentrations. In parallel, corresponding hemoglobin values shall be obtained invasively to form the basis for the development of an algorithm for the device.

To determine inflammation, the frequencies of vasomotion and oxygenation of the tissue are measured non-invasively with the Haemospect®. Various blood parameters for iron and inflammation will also be determined, such as ferritin, hepcidin, transferrin, serum iron, white blood cell count and CRP.

ELIGIBILITY:
Inclusion Criteria:

* all children in treatment for renal insufficiency in FUNDANIER

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects (n ≈ 80) will be enrolled in the Fundación del Niño Enfermo Renal (FUNDANIER) in Guatemala-City. Approximately 50% of the patients in this institution are on hemodialysis and 50% are on peritoneal dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | 1 day
Iron parameters | 1 day
  Serum iron, ferritin, transferrin, transferrin saturation, TIBC, hepcidin
Inflammation parameters | 1 day
  Ferritin, hepcidin, CRP, white blood cell count, ESR

SECONDARY OUTCOMES:
anthropometric data | 1 day
  weight, height, WAZ, HAZ and WHZ